CLINICAL TRIAL: NCT02798510
Title: Clinical Trial of Adjuvant Chemotherapy Followed by Concurrent Chemoradiotherapy Compared With Adjuvant Chemotherapy Alone in Patients With Gallbladder Carcinoma and Extrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhi-Gang Ren, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-PG001
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Malignant Neoplasm Other Gallbladder/Extrahepatic Bile Duct
Keywords: Gallbladder Carcinoma; Extrahepatic Cholangiocarcinoma; Chemoradiotherapy
MeSH Terms: conditions — Gallbladder Neoplasms; Cholangiocarcinoma | interventions — Chemoradiotherapy; Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Patients in arm 1 will receive adjuvant chemotherapy followed by concurrent chemoradiotherapy. Patients will receive four cycles of gemcitabine (1,000mg/m2 intravenously on days 1 and 8) and capecitabine (1,500mg/m2 per day on days 1 to 14) every 21 days followed by concurrent capecitabine (1,330mg/m2 per day) and radiotherapy (50.4Gy/28fx to regional lymphatics with or without tumor bed)
  Interventions: Radiation: Concurrent Chemoradiotherapy; Drug: capecitabine; Drug: gemcitabine
- Arm 2 (Active Comparator): Patients in arm 2 will receive six cycles chemotherapy of gemcitabine (1,000mg/m2 intravenously on days 1 and 8) and capecitabine (1,500mg/m2 per day on days 1 to 14) every 21 days
  Interventions: Drug: capecitabine; Drug: gemcitabine

INTERVENTIONS:
Radiation: Concurrent Chemoradiotherapy
  Arms: Arm 1
Drug: capecitabine
Drug: gemcitabine

SUMMARY:
The present study is designed to determine whether adjuvant concurrent chemoradiotherapy improves overall survivals.

DETAILED DESCRIPTION:
The role of adjuvant radiotherapy in gallbladder carcinoma (GBCA) or extrahepatic cholangiocarcinoma (EHCC) is unknown. A retrospective study suggested that chemoradiotherapy provides greater benefit than chemotherapy alone in GBCA patients. SWOG S0809, a phase II study showed that adjuvant chemoradiotherapy has promising efficacy in GBCA or EHCC. The present phase III clinical trial is designed to compare adjuvant concurrent chemoradiotherapy with chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* The patients with pathologic diagnosis of gallbladder carcinoma (GBCA) or extrahepatic cholangiocarcinoma (EHCC) after radical resection.
* The patients with pathologic stage T2-4 or N1 in R0 resection or positive resection margins (R1).
* Aged 18 to 70 years old, male or female, body condition score generally ECOG 0～2, expected survival ≥ 6 months.
* Subjects were no major organ dysfunction, blood, liver, kidney and heart function was normal, the specific requirements of laboratory indicators:

  * Blood: Absolute neutrophil count > 1.5 × 109 / L, Platelet count > 100 × 109 / L, Hb > 8.0g/dl.
  * Liver function: serum bilirubin less than 1.5 times the upper limit of normal; ALT and AST less than 2.5 times the upper limit of normal.
  * Renal function: creatinine less than 1.5 times the upper limit of normal.
* Patients who can understand the circumstances of this study and signed informed consent.

Exclusion Criteria:

* Pregnancy, breast-feeding patients；
* Patients received prior anticancer therapy for the current malignancy or upper abdominal radiotherapy or chemotherapy at any time.
* Patients with malignant ascites.
* Patients with purulent and chronic infected wounds which delayed healing.
* Patients with liver, kidney and heart failure and coronary heart disease, angina, myocardial infarction, arrhythmia, cerebral thrombosis, stroke and other serious cardiovascular and cerebrovascular disease;
* Patients has a history of mental illness and difficult to control;
* Patients who was considered inappropriate to participate in the trials by the researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
overall survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: zhigang ren, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan university cancer hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Luvira V, Satitkarnmanee E, Pugkhem A, Kietpeerakool C, Lumbiganon P, Pattanittum P. Postoperative adjuvant chemotherapy for resectable cholangiocarcinoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD012814. doi: 10.1002/14651858.CD012814.pub2. PMID 34515993